CLINICAL TRIAL: NCT05214807
Title: Safety and Performance of an Intra-articular Injection of KiOmedine CM-Chitosan in Patients With Advanced Symptomatic Knee Osteoarthritis: Single-blind Randomized Controlled Trial With a 12-month Follow-up Period.
Brief Title: Long-term Safety and Performance of KiOmedine CM-Chitosan Supplementation in Advanced Symptomatic Knee Osteoarthritis
Acronym: PIONEER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kiomed Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KIO014-PIONEER
Record Dates: First submitted 2022-01-17; First posted 2022-01-31 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group receiving Synvisc-One® (Active Comparator)
  Interventions: Device: Synvisc-One®
- IMD group receiving KiOmedine® CM-Chitosan (Experimental)
  Interventions: Device: KiOmedine® CM-Chitosan

INTERVENTIONS:
Device: KiOmedine® CM-Chitosan — KiOmedine® CM-Chitosan is a fluid implant intended for synovial fluid supplementation for the symptomatic treatment of osteoarthritis (OA). This Investigational Medical Device (IMD) is administered via intra-articular injection and is classified as a Class III Device under Council Directive 93/42/EEC (Annex IX, rule 8). A key component of the IMD is a soluble derivative of highly purified chitosan of non-animal origin, an exclusive natural linear glucosamine polysaccharide extracted from the edible white mushroom, Agaricus bisporus. KiOmedine® CM-Chitosan is sterile, non-pyrogenic, resorbable and composed of 2% (w:w) carboxymethyl chitosan (CM-chitosan).
  Arms: IMD group receiving KiOmedine® CM-Chitosan
Device: Synvisc-One® — Synvisc-One (Hylan G-F 20) is a sterile, nonpyrogenic, elastoviscous fluid containing Hylan A and Hylan B polymers produced from chicken combs. Hylans are derivatives of hyaluronan (sodium salt of hyaluronic acid) and consist of repeating disaccharide units of N-acetylglucosamine and sodium glucuronate. Hylan A has an average molecular weight of approximately 6,000,000 daltons and hylan B is a hydrated gel. Hylan G-F 20 contains Hylan A and Hylan B (8.0 mg ± 2.0 mg per ml) in buffered physiological sodium chloride solution (pH 7.2 ± 0.3) and is unique in that the hyaluronan is chemically crosslinked.
  Arms: Control group receiving Synvisc-One®

SUMMARY:
A single-blind randomized controlled design intended for the assessment of safety and performance of a single intra-articular injection of the IMD. In the study, 92 patients meeting eligibility criteria will be randomly assigned to two groups respectively of 46 subjects receiving a single injection of the IMD and 46 subjects receiving a single injection of Synvisc-One® (Hylan G-F 20) which is selected as comparator. Each patient will be blinded for the treatment he/she receives at the injection visit (single blinding).

The patients will be followed for 12 months post-injection to understand long-term safety and performance effects.

The study aims to evaluate the safety and performance of a single injection of KiOmedine® CM-Chitosan compared to the comparator device (Synvisc-One®) in patients with advanced symptomatic knee osteoarthritis.

The non-inferiority hypothesis for the primary performance objective is that the percentage mean reduction in pain from baseline at 6 months in the KiOmedine® CM-Chitosan group is non-inferior to that of the comparator group considering a non-inferiority margin. If the hypothesis of non-inferiority is met, then superiority testing will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 40 years and ≤ 85 years.
* Advanced osteoarthritis, involving one or multiple of the following phenotypes: tricompartmental osteoarthritis, isolated or severe patella-femoral osteoarthritis, a BMI ≥ 30 kg/m2, and/or a Kellgren and Lawrence grade III or IV classification:

  * Patellofemoral osteoarthritis referring to symptoms, including pain, that are principally of patellofemoral origin (Patellar syndrome).
  * Radiological Kellgren and Lawrence grade III to IV from a standing knee radiograph taken less than 6 months previously.
* Symptomatic osteoarthritis diagnosed via radiographic assessment and according to the clinical and radiological criteria of the American College of Rheumatology (ACR).
* Single intra-articular corticosteroid injection during the screening visit (V0), according to standard clinical practice, to resolve clinically apparent knee effusion and/or local signs of inflammation. Patients can only participate in the clinical investigation when there is no sign of effusion and no local signs of inflammation at the patient in visit (V1) which is planned 1-2 weeks after the screening visit.
* Moderate to severe symptomatic pain (i.e., total score on the WOMAC pain subscale ≥12) at screening visit in the treatment knee not or poorly responding to first line non-opioid analgesics and non-steroidal anti-inflammatory drug in oral uptake.
* Pain criteria assessed prior to injection using the 5-point Likert WOMAC pain score:

  * Treatment knee: moderate to severe pain in the most affected knee (i.e., total score on the WOMAC pain subscale ≥12).
  * Non-treatment knee: no to mild pain in the less/non affected knee (i.e., total score on the WOMAC pain subscale ≤5).
* Fully ambulatory patient for functional evaluation.
* For female NOT surgically sterile (tubal ligation or hysterectomy) or NOT postmenopausal for at least one year, must have an effective contraception (pill, patch, ring, diaphragm, implant or intrauterine device).
* Able to understand and follow the instructions of the study.
* Having signed a written informed consent.

Exclusion Criteria:

Meeting one of the following contraindications as stated in the instructions for use of KiOmedine® CM-Chitosan or Synvisc® One:

* A known allergy or hypersensitivity to any of the product components,
* Infections or skin disease at or around the injection site,
* Severe inflammation, synovitis or inflammatory arthritis of the knee joint,
* A history of autoimmune and crystal diseases,
* Evidence of lymphatic or venous stasis or serious blood disorders.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2023-08-20 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
Percentage change from baseline in knee pain at 6 months post-injection measured by the 5-point Likert WOMAC pain scale. | 6 months

SECONDARY OUTCOMES:
Percentage change from baseline in knee pain measured by the 5-point Likert WOMAC pain scale. | 2 weeks, 3 months, 9 months and 12 months post-injection.
Percentage change from baseline in knee stiffness measured by the 5-point Likert WOMAC stiffness scale. | 2 weeks, 3 months, 6 months, 9 months, and 12 months post-injection.
Percentage change from baseline in physical functioning measured by the 5-point Likert WOMAC physical functioning scale. | 2 weeks, 3 months, 6 months, 9 months, and 12 months post-injection.
Percentage change from baseline in the total WOMAC score. | 2 weeks, 3 months, 6 months, 9 months, and 12 months post-injection.
Percentage change from baseline in patient's pain and global assessment using an 11-point numerical rating scale. | 2 weeks, 3 months, 6 months, 9 months, and 12 months post-injection.
Response to treatment according to the Osteoarthritis Research Society International (OARSI) Standing Committee for Clinical Trials Response Criteria Initiative and the Outcome Measures in Rheumatology (OMERACT). | 2 weeks, 3 months, 6 months, 9 months and 12 months post-injection.
Treatment responders with >40% improvement from baseline in pain measured by the 5-point Likert WOMAC pain scale. | 2 weeks, 3 months, 6 months, 9 months, and 12 months post-injection.

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Schifflers, MD, Study Director — Kiomed Pharma
Locations (1):
- Hip and Knee Unit, Ghent, Belgium